CLINICAL TRIAL: NCT07135817
Title: Preoperative Stereotactic Radiotherapy for Treatment of Spinal Metastases
Acronym: PRESTRASM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Rami El Shafie, Principal Investigator, University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/5/24
Record Dates: First submitted 2025-08-01; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Spinal Metastases; Solid Tumor Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Stereotactic Body Radiotherapy + Surgery (Experimental): Participants will receive hypofractionated Stereotactic Body Radiotherapy (SBRT) to spinal metastases in 1-3 fractions within one week after informed consent. SBRT will be planned using MRI co-registered with planning CT and delivered following institutional immobilization standards and ESTRO guidelines. Surgical intervention will follow within a maximum of 10 days after informed consent and includes decompression of the spinal canal and/or dorsal instrumentation, depending on clinical indication.
  Interventions: Radiation: Preoperative Stereotactic Body Radiotherapy (SBRT); Procedure: Spinal Surgery for Decompression and/or Stabilization

INTERVENTIONS:
Radiation: Preoperative Stereotactic Body Radiotherapy (SBRT) — Hypofractionated SBRT delivered in 1-3 fractions within 10 days before surgery, using MRI-based planning and institutional immobilization standards according to ESTRO guidelines.
Procedure: Spinal Surgery for Decompression and/or Stabilization — Surgical intervention is performed following SBRT, based on clinical indication. It includes decompression of the spinal canal in cases of spinal cord or nerve compression (via laminectomy and/or foraminotomy), and/or dorsal instrumentation for unstable spines using pedicle screws guided by a neuronavigation system (Brainlab, Munich, Germany)

SUMMARY:
The goal of this interventional clinical trial is to evaluate the efficacy and safety of preoperative hypofractionated Stereotactic Body Radiotherapy (SBRT) in the treatment of patients undergoing surgery for spinal metastases.

The main questions this study aims to answer are:

* Does preoperative SBRT result in local tumor control at the involved spinal segments as assessed by MRI/CT scan at 3 and 6 months postoperatively?
* What are the postoperative outcomes in terms of pain intensity, functional status and quality of life?

Participants will receive hypofractionated SBRT to spinal metastases shortly before surgical intervention.

Participants will undergo preoperative and follow-up assessments, including:

* MRI and CT scans before and after surgery and at 3 and 6 months after surgery to measure tumor size
* Pain questionnaires where patients rate their current pain, worst pain, and average pain in the last 24 hours on a scale from 0 (no pain) to 10 (worst pain imaginable)
* A short questionnaire (Karnofsky Performance Status) to assess the patient's general ability to carry out daily activities
* Several patient questionnaires to evaluate back pain, physical limitations, and overall quality of life (Oswestry Disability Index, EORTC QLQ-C30, and EORTC QLQ-BM22)

ELIGIBILITY:
Inclusion Criteria:

* Indication for surgical treatment of a spinal tumor
* Age: older or 18 years
* Estimated survival > 6 months
* The patient is able to understand the nature, significance and scope of the clinical study in the context of patient information and to base the decision to participate in the study on this.

Exclusion Criteria:

* Age: < 18 years
* Motor deficit or loss of bladder and bowel control that urges an emergency surgical decompression
* Tumor extent does not allow hypofractioned SBRT (1-3 fractions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Local Tumor Control | 3 months after treatment

SECONDARY OUTCOMES:
Local Tumor Control | 6 months after treatment
Pain relief | at discharge from initial hospitalization (typically within 5-10 days after surgery), 3 and 6 months after treatment
  Pain rating measured by numerical rating scale (zero to ten): This is conducted by asking the patients to rate their 1) present pain, as well as 2) the worst pain they had experienced in the last 24 hours, and 3) the average pain experienced in the last 24 hours on a numeric rating scale (NRS: 0 = "no pain", 10 = "worst pain imaginable").
Wound Healing Complications at Hospital Discharge | at discharge from initial hospitalization (typically within 5-10 days after surgery)
EORTC QLQ-C30 Scores | 3 and 6 months after treatment
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) is a validated 30-item questionnaire to assess cancer patients' general health status and quality of life. Scores range from 0 to 100. For global health and functioning scales, higher scores indicate better outcomes. For symptom scales, higher scores indicate worse symptoms.
EORTC QLQ-BM22 Scores | 3 and 6 months after treatment
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Bone Metastases module (EORTC QLQ-BM22) is a validated 22-item patient-reported outcome measure designed to assess quality of life specifically in patients with bone metastases. It includes functional and symptom domains. Scores range from 0 to 100. Higher scores in symptom scales indicate worse symptoms; higher scores in functional scales indicate better function.
Oswestry Disability Index (ODI) | 3 and 6 months after treatment
  The Oswestry Disability Index (ODI) is a validated patient-reported outcome questionnaire used to assess the degree of disability and functional impairment due to low back pain. It consists of 10 items covering activities of daily living. Scores range from 0% to 100%, with higher scores indicating greater disability.
Number of participants with radiologically confirmed instrumentation failure | 6 months after surgery
  Instrumentation failure will be assessed based on postoperative spinal imaging (CT and MRI). Failure is defined as signs of implant loosening, breakage, displacement, or the need for surgical revision. Imaging will be evaluated by a radiologist according to institutional standards. The number of affected participants will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided